CLINICAL TRIAL: NCT06936215
Title: Safety and Efficacy of Baricitinib on Skin Tightening in Diffuse Cutaneous Systemic Sclerosis: A Comparative Study With Methotrexate
Acronym: BardSSc
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Fahad Hossain, Doctor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5011
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-01

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: Baricitinib in diffuse cutaneous systemic sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — baricitinib; Methotrexate; Folic Acid

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A participants will get tab. baricitinib 4 mg daily
  Interventions: Drug: tab baricitinib 4 mg daily
- Group B (Active Comparator): Group B participants will be given tab. Methotrexate 25 mg weekly with folic acid 5 mg weekly
  Interventions: Drug: tab methotrexate 25 mg weekly with folic acid 5 mg weekly

INTERVENTIONS:
Drug: tab baricitinib 4 mg daily — Group A participants will be given tab. Baricitinib 4 mg daily
  Arms: Group A
Drug: tab methotrexate 25 mg weekly with folic acid 5 mg weekly — group A participants will be given tab. baricitinib 4 mg daily and group B participants will be given tab. methotrexate 25 mg weekly with folic acid 5 mg weekly
  Arms: Group B

SUMMARY:
Systemic sclerosis (SSc) is a systemic autoimmune disease. It causes progressive skin tightening, pulmonary fibrosis, organ damage and many other physical dysfunctions. It is divided into two types, limited cutaneous systemic sclerosis (lcSSc) and diffuse cutaneous systemic sclerosis (dcSSCc). Skin involvement in systemic sclerosis is assessed by modified Rodnan skin score (mRSS). Methotrexate is a drug used in the treatment of skin tightening in SSc but has inconsistent response . Janus kinase (JAK) inhibitors are a class of drugs that may be used in skin involvement in dcSSc. Among them, baricitinib, a JAK 1/2 inhibitor, has shown some efficacy in dcSSc. The aim of this study is to assess the efficacy and safety of baricitinib on skin tightening in dcSSc patients. This open label randomized clinical trial will be conducted in department of rheumatology, BSMMU. Systemic sclerosis will be diagnosed by ACR/EULAR classification criteria 2013. Among them who have diffuse cutaneous involvement will be considered primary entry criteria for this study. Consecutive sampling method will be applied. Participants will be divided into two groups, group A and group B. Group A will be put on tab. baricitinib 4 mg daily and group B will be put on tab. methotrexate 25 mg weekly with folic acid 5 mg weekly. All participants will be assessed for mRSS, CDAI at baseline and laboratory tests like CBC, ESR, CRP, SGPT, serum creatinine, CXR P/A view etc. Follow up will be done at 4, 12, 24 weeks. Response to treatment will be assessed by modified Rodnan skin score. Primary endpoint of efficacy will be assessed by the end of 24th week. adverse effects will be assessed by history, physical examination and investigations. The data will be analyzed by SPSS version 25. results will be recorded using means and standard deviations. Result will be compared among groups with a 95% confidence interval and a p-value 0f<0.05. The degrees of statistical significance between groups will be analyzed by unpaired t test (for quantitative normally distributed data) and Mann Whitney U test for skewed distribution. Qualitative data in between groups will be analyzed by chi square test. Probabilities of association will be assessed by Spearman's rank correlation coefficient. P value of < 0.05 will be regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of diffuse cutaneous systemic sclerosis, as classified using the 2013 American College of Rheumatology

  2. Diffuse cutaneous systemic sclerosis as defined by 2001 LeRoy and Medsger 3. Disease duration ≤ 60 months (defined as time from the first non-Raynaud phenomenon manifestation) 4. mRSS score ≥ 10 at baseline

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Rheumatic disease other than systemic sclerosis. it is acceptable to include patients with fibromyalgia and scleroderma-associated myopathy
2. Limited cutaneous systemic sclerosis or sine scleroderma at the screening visit
3. Major surgery (including joint surgery) within 8 weeks prior to screening visit
4. Any infected ulcer prior to treatment
5. Subjects with any serious bacterial infection (e.g.,chronic pyelonephritis, osteomyelitis, or bronchiectasis) .
6. Oral corticosteroids >10 mg/day of prednisone or equivalent.
7. Mycophenolate mofetil > 2 grams/day prior to baseline
8. Pulmonary disease with FVC ≤ 50% of predicted, or DLCO (uncorrected for hemoglobin) ≤ 40% of predicted
9. Current clinical, radiographic, or laboratory evidence of active TB.
10. Positive for hepatitis B surface antigen at or within 30 days of screening.
11. Positive for hepatitis C antigen at or within 30 days of screening.
12. Current or recent history of uncontrolled clinically significant renal, hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurologic disease.
13. Pregnant or breastfeeding female subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in the protocol for the duration of the study and for at least 28 days after discontinuation of study drug.
14. History of any malignancy in the last 5 years
15. History of SSc Renal Crisis within the 6 months prior to baseline.
16. Patients with a history of anaphylaxis to Baricitinib or methotrexate
17. Any of the following lab results at screening:

    * Hemoglobin <8 g/dl
    * White Blood Cell count <3.0 x 109/L;
    * Absolute Neutrophil count <1.2 x 109/L;
    * Platelet count <100 x 109/L;
    * Absolute Lymphocyte count <0.75 x 109/L.
    * ALT > 3 × the upper limit of normal (ULN) of normal at screening
    * Estimated glomerular filtration rate [GFR] <60mL/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
change in mRSS score | 24 weeks
  mRSS score is recorded at baseline and change in mRSS score is measured in subsequent follow ups at 4, 12 and 24 weeks

SECONDARY OUTCOMES:
Change in CDAI score | 24 weeks
  Baseline clinical disease activity index (CDAI) is recorded and is measured in subsequent follow ups at 4, 12 and 24 weeks
See the side effects of drugs | 24 weeks
  side effect of group A and group B is recorded at 4, 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr MD. Fahad Hossain, MBBS, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- BSMMU, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
participants may not allow sharing all informations with others other than investigator